CLINICAL TRIAL: NCT00747994
Title: Genetic Study of Families Affected by Paget's Disease of Bone
Acronym: PAGET
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Novartis (Industry); Association Rhumatisme et Travail (Unknown)
Responsible Party: Yannick Vacher, Department Clinical Research of Developpement
Other Study IDs: P070203
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: Paget's Disease of Bone
Keywords: Paget's disease of bone; Relatives; Mutations screening; Haplotypes analysis; Linkage analysis; < 55 years; 4 > or = WAFFECTED Bones; bone deformity
MeSH Terms: conditions — Osteitis Deformans

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — collection of extracted DNA, RNA and serum samples and urinary samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
Paget's disease of bone is a frequent bone disorder which usually starts after the age of 40 and which is characterized by bone pain and deformities. Although often without any symptoms, this disease may have severe complications such as fissures, fractures, neurological compression, or deafness. In some cases, it is a genetic disorder transmitted with a dominant autosomal pattern of inheritance: one of the two parents carrying the disease transmits it to his offspring with a risk of 50% for each child. Since 2002, the first gene involved in Paget's disease of bone is known and 14 mutations of this gene have been published. A study confirmed that the presence of those mutations was associated with younger age of onset and more extensive disease. Thus, the knowledge of those genetic factors in the relatives of an affected individual allows the screening of the patients with a higher risk for complications, who may benefit from a medical follow up and earlier treatment, in order to avoid complications. Indeed, Paget's disease of bone may be treated efficiently by bisphosphonates.

This project aims at identifying and collecting over one year, 15 affected individuals affected by Paget's disease of bone and the relatives up to the second degree of relativeness (a total of 100 individuals is expected). The blood samples may be analysed in order to search for mutations of the previously known gene and/or to search for new mutations on new genes.

DETAILED DESCRIPTION:
Background : Paget's disease of bone is a chronic bone disorder with a late onset, usually after the age of 40. This disease is transmitted on a dominant autosomal pattern of inheritance with incomplete penetrance. Since 2002, the first gene (SEQUESTOSOME 1 or SQSTM1) involved in Paget's disease of bone is known. Actually, 14 mutations of this gene located in exons 7 and 8 have been reported in familial forms of the disease as well as in sporadic forms. Although the size of the samples studied in the literature are rather small to establish phenotype genotype correlations, it seems that the presence of those mutations are associated with an earlier onset of the disease and a more extensive disease. However, the presence of those mutations seems not sufficient to explain the whole development of the disease, but functional analyses may help to understand the real effect of those mutations. The link between the genetics and the observation of PARANYXOVIRAL inclusions in the nucleus of osteoclasts is not actually established. The hypothesis of an interaction between gene and environment may be plausible for several authors.

The results of a study on 94 sporadic French patients with Paget's disease of bone lead to the identification of two new mutations of SQSTM1 gene and showed the presence of double SQSTM1 mutations. This study established phenotype genotype correlations, affected individuals who carry a mutation have a younger age at diagnosis and a polyostotic involvement. This phenotype genotype correlation is a major element that may help to target the relatives at risk for complications, who may benefit from an earlier treatment to prevent complications occurrence.

Primary objective : to recruit 15 patients affected by Paget's disease of bone, with a familial form, and their relatives healthy or affected, up to the second degree of relativeness (total of about 100 individuals) for a genetic study on Paget's disease of bone with : DNA collection, blood puncture for RNA collection, serum collection and urinary collection to study the bone remodelling parameters. DNA samples will be used to search for mutations involved in Paget's disease of bone in collaboration with the research center of the University hospital center of LAVAL, Quebec, Canada.

Inclusion and exclusion criteria are described elsewhere.

Description of the protocol:

- Identification of the affected patients (15 index cases). Inclusion visit for the index case : information on the project and signature of the consent, validation of the inclusion criteria for the index case, clinical exam, answers to the questionnaire. Detailed family pedigree and information given to the index case for the relatives up the second degree of relativeness for participation in the present study. Blood puncture and urinary collection, imaging is required in the next three months only if not previously done.

Inclusion visit for the relative, healthy or affected by Paget's disease of bone: Information on the project and signature of the consent, validation of the inclusion criteria, clinical exam and answer to the questionnaire, blood and urinary collection. Imaging is required only for healthy relatives with bone scintigraphy in the next three months or skull and pelvis radiographies. For the affected relatives, imaging tests are required only when not previously done.

Exams realized on the patient for the study:

Each individual, healthy or affected by Paget's disease of bone, included in this study, has to undergo biological tests (alkalies phosphatases, creatinin and gammaGT) and imaging tests if not realized during the past 10 years (bone scintigraphy and /or radiographies of the skull and pelvis). Blood puncture will be done to extract DNA, RNA and serum samples and urinary samples will be collected.

Benefits and risks :

Benefits : The realisation of biological and imaging exams to search for asymptomatic lesions of Paget's disease of bone, may lead to fortuitously identify bone lesions of various etiologies, which treatment and follow up may be beneficial to the relatives, but the kind of benefit is not certain. The identification of a SQSTM1 mutation in a relative may lead to an earlier treatment that may prevent the occurrence of complications. Indeed, there is an efficient medical treatment for Paget's disease of bone (bisphosphonates). There is no benefit for the index case, nor for the affected relatives.

Known risks : Pain due to veinous blood puncture et irradiation with the bone scintigraphy and/or radiographies.

Numbers of patients : 15 patients affected by Paget's disease of bone and their relatives at the first or second degree of relativeness, in a total of about 100 individuals. This number is based on the feasibility of the recruitment and on the fact that those families may be pooled for the analysis with families from Quebec and will allow to increase the power to detect by linkage analysis new mutations, new haplotypes and/or new genes.

Main objective : New mutations or new haplotypes of already identified mutations, new mutations of new genes of the disease.

Expected results :

* According to the frequency of the SQSTM1 mutations in familial forms of the disease, a mutation in this gene may be identified in 1/3 of the families, ie about 5 families. In those families, the haplotypes study may show two major haplotypes containing the P392L mutation. This family material with identified mutation may be useful to search for phenotype genotype correlation and to search for modifier factors (genetic, epigenetic, environmental).
* In the 10 other families, no SQSTM1 mutations are expected. Those families may be pooled to families with the genetic background (French Canadian), who may allow to reach a sufficient power to detect by linkage analysis new regions of the genome that may contain an other gene of Paget's disease of bone.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years,
* patient who underwent a clinical examination,
* patient who gave its written consent,

  1. Each individual (index case) affected by Paget's disease of bone (with diagnosis confirmed by alkalies phosphatases analysis and/or imaging with bone scintigraphy and radiographies on the affected sites with a typical aspect of the disease), and :

     * At least one relative affected by Paget's disease of bone with confirmed diagnosis (see above),
     * Or an age at diagnosis < 55 years,
     * Or a polyostotic involvement with at least 4 affected bones,
     * Or the presence of a bone deformity at the time of the diagnosis.
  2. Each relative with established phenotype by imaging (bone scintigraphy and/or radiographies), at first or second degree of relativeness of an index case defined in (a).

Exclusion Criteria:

* Index case with not confirmed Paget's disease of bone by biological and/or radiological examinations,
* Index with confirmed Paget's disease but without relative with the same disease, with an age at diagnosis >55 years, with a number of affected bones <4, without any bone deformity at the time of the diagnosis
* Healthy relatives of a Paget patient who refuse to undergo bone scintigraphy and bone radiographies.
* Individuals < 18 years
* Pregnant or breast
* feeding woman-individual living ina sanitary or social establishment
* individual under guardianship
* individual in an emergency situation
* individual unable to give his consent
* incarcerated individual
* patient not covered by healthcare institutions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 15 patients affected by Paget's disease of bone and their relatives at the first or second degree of relativeness total of about 100 individuals
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To identify new mutations or new haplotypes of mutations already identified, and/or to identify new mutations in new genes of Paget's disease of bone. | 2007-2008

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia Michou, MD PhD, Study Director — CHU Lariboisière
Locations (1):
- CHU Lariboisière, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Collet C, Michou L, Audran M, Chasseigneaux S, Hilliquin P, Bardin T, Lemaire I, Cornelis F, Launay JM, Orcel P, Laplanche JL. Paget's disease of bone in the French population: novel SQSTM1 mutations, functional analysis, and genotype-phenotype correlations. J Bone Miner Res. 2007 Feb;22(2):310-7. doi: 10.1359/jbmr.061106. PMID 17129171
- [Background] Morissette J, Laurin N, Brown JP. Sequestosome 1: mutation frequencies, haplotypes, and phenotypes in familial Paget's disease of bone. J Bone Miner Res. 2006 Dec;21 Suppl 2:P38-44. doi: 10.1359/jbmr.06s207. PMID 17229007